CLINICAL TRIAL: NCT01609517
Title: The Influence of Body-mass Index on the Outcome of Spinal Anesthesia for Total Knee Replacement Arthroplasty
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sangmin M. Lee, Professor, Samsung Medical Center
Other Study IDs: 2012-04-089-001
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Spinal Anesthesia; Success or Failure of Spinal Anesthesia
Keywords: Spinal anesthesia; determinant; duration
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese group: patients with BMI >= 30.0 kg/m2 who received spinal anesthesia with heavy marcaine
  Interventions: Drug: Spinal anesthesia (heavy bupivacaine)
- Non-obese group: patients with BMI < 30.0 kg/m2 who received spinal anesthesia with heavy marcaine
  Interventions: Drug: Spinal anesthesia (heavy bupivacaine)

INTERVENTIONS:
Drug: Spinal anesthesia (heavy bupivacaine) — Spinal anesthesia with heavy bupivacaine of 6, 7, 8, 9, 10, 11 mg
  Other Names: Spinal anesthesia; heavy bupivacaine

SUMMARY:
In these prospective observational study, the investigators are trying to evaluate (1) the influence of body-mass index on spinal anesthetic outcome and (2) the determinants on spinal anesthetic outcome by logistic regression analysis.

DETAILED DESCRIPTION:
Although the spread of spinal anesthetic drug is unpredictable, patients factors (age, gender, height,weight, body-mass index), spinal anatomy, anesthetic drug dose, and lumbosacral cerebrospinal fluid volume are known to be the determinants of sensory block level. Among these determinants, the influence of body-mass index (BMI) on spinal anesthesia is controversial, and there is no specific guideline showing the relative priority of these determinants.

Therefore, in these prospective observational study, the investigators are trying to evaluate (1) the influence of body-mass index on spinal anesthetic outcome and (2) the relative influence of these determinants on spinal anesthetic outcome by logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing spinal anesthesia in Samsung Medical Center during study period
* American Society of Anesthesiologist Physical Status classification I ~ III

Exclusion Criteria:

* Bupivacaine allergy
* medical history of spinal surgery
* Diabetic neuropathy
* active infection at the lumbosacral area
* other contraindication of spinal anesthesia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing spinal anesthesia in Samsung Medical Center during study period
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
spinal anesthetic success/ failure | at 2 hour after the anesthetic induction
  when (1) a bilateral T12 sensory block to pinprick within 15 minutes of intrathecal drug administration with sensory/motor block scale ≥ 2 and (2) the level of sensory block at the end of surgery was higher than or equal to T12 with sensory/motor block scale ≥ 2.

SECONDARY OUTCOMES:
Peak level of sensory block at anesthesia induction | during 20 min after anesthetic induction
  Sensory block levels determined by pinprick test
Spinal anesthesia sensory/motor block level at the end of surgery | 2 hours after induction (at the end of surgery)
  Spinal anesthesia block level as determined by Pinprick sensory test with Bromage scale.
  Sensory 0 = an ability to appreciate a pinprick as sharp; 1 = perception of a pinprick as less sharp than in unblocked areas; 2 = perception of a pinprick as touch but not sharp (analgesia); 3 = an inability to feel pinprick(anesthesia).
  Bromage Scale 0 = ability to lift an extended knee at the hip; 1 = ability to flex the knee but not to lift an extended leg; 2 = ability to flex toes only; 3 = inability to move.
the incidence of tourniquet pain | at 90 min afer anesthetic induction
  the incidence of tourniquet pain during the tourniquet time reported by the patient (NRS >= 2)
Incidence of hypotension, bradycardia | during 2 hours after anesthesia induction
  Incidence of hypotension, bradycardia total dose of ephedrine Lowest mean blood pressure Incidence of vomiting, shivering

CONTACTS AND LOCATIONS:
Overall Officials: Sangmin M. Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Ji Sun Hahm, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea